CLINICAL TRIAL: NCT00284362
Title: Prospective and Comparative Analysis of Arthroscopic and Open Surgery for Hallux Rigidus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/095
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Hallux Rigidus
MeSH Terms: conditions — Hallux Rigidus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Arthroscopic or open surgery for hallux rigidus

SUMMARY:
Comparison between arthroscopic and open surgery for hallux rigidus.

ELIGIBILITY:
Inclusion Criteria:

* Hallux rigidus

Exclusion Criteria:

-

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalisation
Duration of rehabilitation and sick leave
Wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be